CLINICAL TRIAL: NCT05217147
Title: An Investigation of Clinical Parameters and Biomarkers Associated With Angiogenesis, Proliferation, Cell Adhesion and Invasion in Laryngeal Carcinoma
Brief Title: An Investigation of Biomarker Candidate Molecules in Laryngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gurcan GUNAYDIN, MD, PhD, Associate Professor, Hacettepe University
Other Study IDs: THD-2019-18414
Record Dates: First submitted 2022-01-04; First posted 2022-02-01 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-01

CONDITIONS: Larynx Cancer; Larynx Carcinoma
Keywords: larynx carcinoma; angiogenin; endoglin; vegf; svegfr-1; vegfr-2; osteoponitn; biomarker
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: 60 patients with laryngeal carcinoma
  Interventions: Other: Obtaining blood samples
- Control group: 20 healthy age- and sex- matched controls
  Interventions: Other: Obtaining blood samples

INTERVENTIONS:
Other: Obtaining blood samples — Blood samples were obtained at time of diagnosis and will be analyzed for the levels of biomarker candidate molecules.

SUMMARY:
The aim of this study was to determine serum levels of VEGF, sVEGFR1, VEGFR2, IGFBP-3, angiogenin and endoglin in patients with larynx squamous cell carcinoma; investigate their association with clinical parameters and determine their diagnostic and prognostic value.

DETAILED DESCRIPTION:
Although there has been a significant increase in survival in many other cancer types through the years, no significant increase has been achieved in laryngeal SCC survival rates in the last 50 years. Despite the advancements in surgical techniques, organ preservation protocols and multidisciplinary approach, significant amount of patients have been living with morbidity or dying due to recurrence and metastasis. This lack of significant improvement in mortality rates creates the need for reliable and accurate biomarkers in early diagnosis, treatment and follow-up. Considering that the prognosis of two patients at the same clinical stage and treated with the same treatment protocol may differ, it suggests that there may be some differences at the molecular level apart from clinical stages.

This study was mainly prepared to determine serum levels of VEGF, sVEGFR1, VEGFR2, IGFBP-3, angiogenin and endoglin in patients with larynx squamous cell carcinoma; investigate their association with clinical parameters and determine their diagnostic and prognostic value.

To reach these aims, 60 patients who were prospectively and consecutively recruited from those who admitted to Hacettepe University, Department of Otorhinolaryngology, Ankara, Turkey, and were diagnosed with LSCC between May 2018 and February 2020. 20 healthy and age-matched controls were chosen from the hospital staff and relatives of the patients. Serum samples were obtained from all participants at the time of diagnosis, centrifuged and stored at -80 C. ELISA method will be used to analyze the serum levels of VEGF, sVEGFR1, VEGFR2, IGFBP-3, angiogenin and endoglin.

Data analysis will reveal if there are any association between biomarker candidate molecules and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* 60 male or female patients with a newly diagnosed laryngeal squamous cell carcinoma
* Patients without any previous history of laryngeal carcinoma
* 20 healthy, age- and sex- matched controls

Exclusion Criteria:

* Previous history of laryngeal squamous cell carcinoma
* Having comorbid systemic diseases like DM, hypertension, cardiologic or rheumatologic diseases
* Having malign tumors elsewhere
* History of chemotherapy/radiotherapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included 60 patients who were prospectively and consecutively recruited from those who admitted to Hacettepe University, Department of Otorhinolaryngology, Ankara, Turkey. 20 healthy and age-matched controls were chosen from the hospital staff and relatives of the patients.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Serum levels of biomarker candidate molecules | Basal
  Serum levels of:
  VEGF in pg/ml
  sVEGFR1 in pg/ml
  VEGFR2 in pg/ml
  IGFBP-3 in pg/ml
  angiogenin in pg/ml
  and endoglin in pg/ml
  will be determined in all participants
Stage | Basal
  Disease stage as stage as early (I-II) or late (III-IV)
Diagnostic sensitivity and specifity of biomarker candidate molecules | Basal
  Receiver operating characteristic analysis will be performed to determine a significant level of any biomarker candidate molecules for diagnostic sensitivity and sensitivity.
  Sensitivity and specifity as percentages (%)
Tumor grade | Basal
  Tumor grade as poor, moderate or well
Recurrence status | 18 months after reaching the target patient number
  Recurrence status as yer or no
Tumor localization | Basal
  Tumor localization as glottic/supraglottic or transglottic
Treatment modality | Basal
  Treatment modality as surgical, non-surgical or combined

SECONDARY OUTCOMES:
Survival analysis parameters | 18 months after reaching the target patient number
  All the patients were contacted for survival analysis.
  Overall and disease-free survival will be measured in months and survival rates will be calculated in percentages (%).
  Overall survival and disease-free survival rates will be calculated according to levels of biomarker candidate molecules and assessed for any association with any molecule.

CONTACTS AND LOCATIONS:
Overall Officials: Gurcan Gunaydin, MD, PhD, Principal Investigator — Hacettepe University Cancer Institute; Nilda Suslu, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University Cancer Institute, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No